CLINICAL TRIAL: NCT06075498
Title: Comparison of Analgesia Efficacy of Transversus Abdominis Plane Block and Posterior Approach Quadratus Lumborum Block After Open Radical Retropubic Prostatectomy Operation
Brief Title: Comparison of Analgesia Efficacy of Transversus Abdominis Plane Block and Posterior Approach Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Eylem Yaşar, Specialist, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 22/III
Record Dates: First submitted 2022-01-24; First posted 2023-10-10 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Acute Post-operative Pain; Nerve Block; Prostate Cancer
Keywords: quadratus lumborum block, transversus abdominis plane block
MeSH Terms: conditions — Pain, Postoperative; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: patients who underwent open retropubic prostatectomy
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Postoperative follow-up was evaluated by a research assistant blind to the procedure.
  groups 1 and 2 were presented to the Outcome Assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plane block (Active Comparator): The group that underwent bilateral transversus abdominis plane block with 0.375 mg 20 ml bupivacaine on each side after open retropubic prostatectomy operations
  Interventions: Procedure: transversus abdominis plane block,
- quadratus lumborum plane block (Active Comparator): The group that underwent bilateral quadratus lumborum plane block with 0.375 mg 20 ml bupivacaine on each side after open retropubic prostatectomy operations
  Interventions: Procedure: transversus abdominis plane block,

INTERVENTIONS:
Procedure: transversus abdominis plane block, — 2 different plan blocks; 1. transversus plane block 2. quadratus lumborum plane block
  Other Names: quadratus lumborum plane block

SUMMARY:
Prostate cancer is the second most common cancer and the fifth in cancer-related deaths. Open radical retropubic prostatectomy is the most common surgical treatment for localized prostate cancer. Open radical retropubic prostatectomy is associated with moderate pain. Severe pain in the postoperative period affects the length of hospital stay and morbidity. Multimodal analgesia applications for the management of postoperative pain are the main component of post-surgical recovery. Different analgesia modalities, including systemic opioid use and neuraxial analgesia, have been used for pain control after retropubic radical prostatectomy. Side effects of systemic and intrathecal opioids limit the potential benefits of these agents. Transversus abdominis plane block and quadratus lumborum block are blocks that can be used for postoperative analgesia in the abdominal and pelvic regions. There is no study in the literature comparing the efficacy of these two blocks for postoperative analgesia in open radical retropubic prostatectomy and their effects on narcotic consumption.

DETAILED DESCRIPTION:
Scope: Open radical retropubic prostatectomy operation is associated with moderate postoperative pain and affects hospital stay and morbidity. Nerve blocks used for postoperative analgesia are one of the components of multimodal analgesia.

Transversus abdominis plane block (TAP) is a regional block (T7-L1) that blocks the sensory afferents of the anterior abdominal wall. It was first introduced as an anatomical landmark-based technique through Petit's lumbar triangle. Since then, the ultrasound-guided block technique has been defined and the effectiveness of this block in postoperative pain control in abdominal and gynecological surgeries has been demonstrated. The sensory distribution of TAP block includes the incisional pain of open prostatectomy. TAP block technique has been shown to be a safe and effective method of postoperative analgesia in various general surgery, urological surgery, plastic surgery and pediatric surgery operations. In addition, postoperative pain management after lower abdominal surgeries has been recommended as part of ERAS protocols.

Quadratus lumborum block (QL) is used as one of the postoperative pain methods after abdominal surgery in all age groups. It has been reported that QL block with a posterior approach extends more easily into the thoracic paravertebral space or the thoracolumbar plane and can create analgesia from T 7 to L 1. The use of posterior QL (QL-2) blocks for postoperative analgesia after open retropubic prostatectomy operations has not been studied before and it is not known which one is superior.

The primary aim of this study was to compare the analgesic efficacy of transversus abdominis plane block and posterior approach quadratus lumborum block and opioid consumption within 24 hours postoperatively. The secondary aim is to determine whether there is a difference in terms of time to first analgesic consumption, duration of sensory block, opioid-related side effects (postoperative nausea and vomiting, itching, sedation), patient satisfaction, and complications related to the block.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-II patients who can adapt to the pain assessment scale will be included in the study.

Exclusion Criteria:

* Patients under 18 years of age
* ASA IV patients
* patients with known allergy to analgesic drugs
* patients with any contraindications for the regional technique (patients with coagulation disorders, injection site infection, patients allergic to local anesthetics)
* patients with chronic analgesic use
* body mass patients with an index over 35 kg/m2

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients will be included in the study, as there are patients who underwent prostate surgery.
Enrollment: 66 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
To compare the two groups analgesic efficacy and opioid consumption within 24 hours postoperatively. | 24 hours postoperatively
  Comparing the analgesic effectiveness of the transversus abdominis plane block and posterior approach quadratus lumborum block and opioid intake and patient pain within 24 hours after surgery

SECONDARY OUTCOMES:
Duration of sensory block, opioid-related side effects (postoperative nausea and vomiting, itching, sedation), patient satisfaction and complications related to the block. | 24 hours postoperatively
  To determine whether there is a difference in terms of time until the first analgesic consumption, duration of sensory block, opioid-related side effects (postoperative nausea and vomiting, itching, sedation), patient satisfaction and complications related to the block.

CONTACTS AND LOCATIONS:
Overall Officials: basak altiparmak, Study Chair — Mugla Sitki Kocman University Department of Anesthesia; ahmet pinarbasi, Study Chair — Mugla Sitki Kocman University Department of Anesthesia; ilker akarken, Study Chair — Mugla sitki kocman department of urology; bakiye ugur, Study Chair — Mugla Sitki Kocman Universty of Anaesthesia; eylem yasar, Principal Investigator — Mugla Sitkı Kocman Training and research hospital
Locations (1):
- Mugla Sitki Kocman Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only the IPD (after the unidentification of the patients) will be available by correspondence author e-mail.